CLINICAL TRIAL: NCT00237783
Title: Hemodynamic Changes During Dialysate Sodium Individualization in Hemodialysis Patients
Brief Title: Safety of Dialysate Sodium Individualization in Hemodialysis Patients With Intradialytic Hypotension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit enough subjects
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP0008
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hemodialysis; Hypotension
Keywords: Renal dialysis; Hypotension; Dialysis solutions
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dialysate sodium (140 mmol/L) (Active Comparator): dialysate sodium (140 mmol/L)
  Interventions: Drug: dialysate sodium (140 mmol/L)
- individualized dialysate sodium (Experimental): individualized dialysate sodium (same concentration as the average pre-HD serum sodium during the baseline period)
  Interventions: Drug: individualized dialysate sodium

INTERVENTIONS:
Drug: dialysate sodium (140 mmol/L)
  Arms: standard dialysate sodium (140 mmol/L)
Drug: individualized dialysate sodium — individualized dialysate sodium (same concentration as the average pre-HD serum sodium during the baseline period)
  Arms: individualized dialysate sodium

SUMMARY:
Low blood pressure (hypotension) during dialysis afflicts approximately 25% of hemodialysis patients. In this pilot study, we will evaluate the safety and effects of individualizing the sodium concentration in the dialysate according to the patient's own plasma sodium levels. We hypothesize that patients will have less thirst and less weight gain during the intervention leading to easier fluid removal and less episodes of hypotension.

DETAILED DESCRIPTION:
Hypertension and intradialytic hypotension are common complications in patients on chronic maintenance hemodialysis (HD). Sodium balance is important in mediating both processes. Recent evidence shows that individualization of the sodium concentration in the dialysate to match the patient's own serum sodium results in less thirst, less interdialytic weight gain, less HD-related symptoms, and better blood pressure control. In this project we plan to evaluate the safety and tolerability of sodium individualization in hypotension-prone patients in order to generate pilot data for a larger study in patients with intradialytic hypotension. In this protocol, we will recruit 7 hypotension-prone subjects. We will use an open-label cross-over design with randomized blocks. After a 3-week baseline period where pre-HD serum sodium will be measured weekly to establish each patient's average serum sodium, subjects will be randomized to 2 weeks on standard dialysate sodium (140 mmol/L) or individualized dialysate sodium (same concentration as the average pre-HD serum sodium during the baseline period), then crossed over to the other for another 2 weeks (total study period 7 weeks, 2 weeks baseline, 4 weeks intervention). The remainder of the dialysis prescription, prescribed dry weight and vasoactive drugs will remain unchanged throughout the study. Clinical information, pre/intra/post-HD blood pressure and hemodynamics (cardiac output and systemic vascular resistance), and the frequency and severity of intradialytic symptoms related to hypotension will be collected on HD sessions during the 4 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with intradialytic hypotension

Exclusion Criteria:

* Atrial fibrillation
* Bilateral upper extremity arteriovenous access
* Average plasma sodium >139

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Intradialytic BP change | from study onset through intervention, week 7

SECONDARY OUTCOMES:
Intradialytic changes in cardiac output and peripheral vascular resistance | from study onset through intervention, week 7
Interdialytic weight gain change | from study onset through intervention, week 7
Thirst scores | from study onset through intervention, week 7

CONTACTS AND LOCATIONS:
Overall Officials: Aldo J Peixoto, MD, Principal Investigator — Yale University and VA Connecitcut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] de Paula FM, Peixoto AJ, Pinto LV, Dorigo D, Patricio PJ, Santos SF. Clinical consequences of an individualized dialysate sodium prescription in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1232-8. doi: 10.1111/j.1523-1755.2004.00876.x. PMID 15327422